CLINICAL TRIAL: NCT03380221
Title: Effects of Fresh Watermelon Consumption on Satiety and Cardiometabolic Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HS-2017-0139
Record Dates: First submitted 2017-12-11; First posted 2017-12-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Satiety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Watermelon (Experimental)
  Interventions: Other: Watermelon
- Low fat cookies (Active Comparator)
  Interventions: Other: Low fat cookies

INTERVENTIONS:
Other: Watermelon — Participants will consume 100 Kcal of watermelon fruit (2 cups) daily for 4 weeks.
  Arms: Watermelon
Other: Low fat cookies — Participants will consume 100 Kcal of low fat cookies daily for 4 weeks.
  Arms: Low fat cookies

SUMMARY:
The goal of the proposed study is to determine the effects of fresh watermelon fruit consumption on satiety, metabolic parameters and weight management.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years old
* BMI 25-40

Exclusion Criteria:

* Smoker
* Pregnant woman
* Required dietary supplement use
* Required medication of metabolic disorders
* Allergy to watermelon or gluten

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2028-12-15 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of Satiety | 0, 20, 40, 60, 90 and 120 minutes post snack consumption
  Hunger feeling (appetite) will be examined using visual analog scale (0-10): 0 is least and 10 greatest.

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise and Nutritional Sciences, SDSU, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lum T, Connolly M, Marx A, Beidler J, Hooshmand S, Kern M, Liu C, Hong MY. Effects of Fresh Watermelon Consumption on the Acute Satiety Response and Cardiometabolic Risk Factors in Overweight and Obese Adults. Nutrients. 2019 Mar 12;11(3):595. doi: 10.3390/nu11030595. PMID 30870970